CLINICAL TRIAL: NCT00192309
Title: A Randomized, Open-Label, Placebo-Controlled Trial to Investigate the Kinetics of the Immune Responses Elicited by a Liquid Formulation of Influenza Virus Vaccine, Trivalent,Types A & B, Live, Cold-Adapted (CAIV-T) in Healthy Adults Aged 18 to <65 Years.
Brief Title: Phase II Study to Investigate the Kinetics of the Immune Response Generated by Influenza Virus Vaccine.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Raburn Mallory, MD/ Sr Dir Clinical Development, MedImmune
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: D153 P004
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — FluMist; Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cold-adapted influenza vaccine (CAIVT) (Experimental): A single intranasal dose of 10^7 fluorescent focus units.
  Interventions: Biological: CAIV-T
- Trivalent inactivated vaccine (TIV) (Active Comparator): A single dose of commercially available Flushield was administered intramuscularly.
  Interventions: Biological: TIV
- Placebo (Placebo Comparator): The 0.2 mL administered intranasally.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CAIV-T — Liquid CAIV-T vaccine for this study consisted of three cold-adapted, attenuated, reassortant strains representing the hemagglutinin (HA) and neuraminidase (NA) antigens of the A/New Caledonia/20/99 (H1N1), A/Panama/2007/99 (H3N2) and B/Yamanashi/166/98 influenza virus strains. The reassortant vaccine strains were grown in specific pathogen-free (SPF) eggs and the allantoic fluid, which contained virus, was harvested, concentrated and purified. Each dose of CAIV-T used in this study was formulated to contain approximately 107 FFU of each of the 6:2 influenza reassortant vaccine strains.
  Other Names: FluMist
  Arms: Cold-adapted influenza vaccine (CAIVT)
Biological: TIV — TIV in this study consisted of Flushield™, manufactured by Wyeth Vaccines, Marietta, PA, USA. Each 0.5 mL dose contained no less than 15 ug of the hemagglutinin antigens from each of the A/New Caledonia/20/99 (H1N1), A/Panama/2007/99 (H3N2), and B/Yamanashi/166/98 strains, making TIV in this study antigenically matched to the influenza strains contained in CAIV-T.
  Other Names: Flushield
  Arms: Trivalent inactivated vaccine (TIV)
Biological: Placebo — Placebo in this study consisted of physiological saline. The total volume of 0.2 mL was administered intranasally with a spray applicator (approximately 0.1 mL into each nostril).
  Arms: Placebo

SUMMARY:
The primary objective of this study was to perform a variety of assays on blood, serum, nasal wash and cell samples obtained from healthy adult subjects for the purposes of developing assays for application in the further investigation of immune responses generated by influenza virus vaccine, trivalent, types A & B, live, cold-adapted (liquid formulation CAIV-T; Wyeth, Marietta, PA).

DETAILED DESCRIPTION:
This was a randomized, open-label, placebo-controlled, outpatient study carried out in healthy adults 18 to < 65 years of age. The study was designed to evaluate the kinetics of the immune responses generated by each of the study products in order to determine the best sampling time for future studies. Subjects were randomized in a 1:1:1 ratio to receive a single dose of either CAIV-T, inactivated influenza virus vaccine (TIV), or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subjects had to have been at least 18 years of age and less than 65 years of age at the time informed consent was obtained;
* Women of child-bearing potential had to use reliable methods of hormonal and/or nonhormonal contraception (which includes cervical cap, diaphragm, condoms with spermicide or IUD) during sexual intercourse throughout the entire study period; a negative urine pregnancy test (with detection limit of less than or equal to 25mIU/mL) no more than 24 hours prior to vaccine administration; and agreed to avoid pregnancy during participation in the study. A urine pregnancy test was also conducted at the completion of study participation. Females who were surgically sterile at time of enrollment were not required to undergo pregnancy testing.
* who were determined by medical history, physical examination and clinical judgement to be eligible for the study.
* who provided written informed consent after the nature of the study has been explained;
* who were available for one month duration of the trial (from enrollment to study completion);
* who could be reached by study staff for the post-vaccination contact [telephone, clinic or home visit].

Exclusion Criteria:

* who were perceived to be unavailable or difficult to contact for evaluation or study visits during the study period;
* with a known or suspected disease of the immune system or those receiving immunosuppressive therapy, including systemic corticosteroids and intranasal steroids; or cytotoxic agents;
* who had an immunosuppressed or an immunocompromised individual living in the same household;
* who had a documented history of hypersensitivity to egg or egg protein or any other component of the study vaccine or placebo;
* who received any commercially-available or investigational injected influenza vaccine in the 6 months prior to enrollment, or a non-study influenza vaccine since enrollment;
* who previously received an intranasally administered influenza vaccine;
* who had any medical conditions that, in the opinion of the investigator, might interfere with interpretation of the study results;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2001-09; Primary Completion 2001-12 (Actual); Study Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
Kinetics of the hemagglutination inhibition antibody response to each vaccine strain | Day 0-28
  The geometric mean titers for each strain between Day 0 and 28 were examined.

SECONDARY OUTCOMES:
Expression of IgA in nasal wash and saliva swab samples | Days 0-28
  Nasal wash and saliva swab IgA antibody titers were expressed as the ratio of specific to total IgA.
Expression of B-cells in peripheral blood | Days 0-28
  The B-cell ELISPOT assays are designed to detect B-cells in the peripheral blood that are actively secreting influenza strain-specific IgG or IgA antibody.
Number of CD3+ peripheral blood mononuclear cells secreting interferon gamma | Days 0-28
  The number of CD3+ peripheral blood mononuclear cells (PBMCs), i.e., T-cells, secreting IFN-γ prior to and after vaccination following in vitro stimulation of these cells using the IFN-γ ELISPOT assay.
Number of subjects with local reactions | Days 0-7
  Local injection site reactions were collected from subjects in the TIV treatment group only.
Number of subjects with systemic reactions | Days 0-7
  Each study subject collected prompted reactogenicity events on a diary card worksheet for 7 days (study days 0 - 6) following vaccination.
Number of subjects with adverse events | Days 0-7
  An Adverse Event (or Adverse Experience, AE) was any untoward, undesired or unexpected clinical event in the form of signs, symptoms, disease or laboratory or physiological observations occurring (in a human being) in a temporal relationship to the use of a WLV product, regardless of causal relationship.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Walker, MD, Principal Investigator — MedImmune LLC
Locations (1):
- David M. Radin, MD, Stamford, Connecticut, United States